CLINICAL TRIAL: NCT03265366
Title: Diagnostic Value of MRI for Allergic Broncho-Pulmonary Aspergilloses
Acronym: ABPA-MR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2016/12
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Allergic Bronchopulmonary Aspergilloses
Keywords: Ultrashort echo time magnetic resonance imaging
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — Tomography, X-Ray Computed; Reference Standards

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABPA (Experimental): 15 patients with ABPA
  Interventions: Device: MRI; Device: CT scan (standard reference)
- Severe asthma (Active Comparator): 12 patients with severe asthma
  Interventions: Device: MRI; Device: CT scan (standard reference)

INTERVENTIONS:
Device: MRI — It will be performed on a 1.5-Tesla MR scanner (MAGNETOM Avanto, Siemens Healthcare, Erlangen, Germany), without injection or inhalation of contrast agent.
Device: CT scan (standard reference) — It will be performed on a 16 (Sensation 16, Siemens®) or 64 channels (Definition 64, Siemens®), without contrast agent injection.

SUMMARY:
The aim of the study is to compare the concordance between chest computerized tomography-scan (CTscan) and Magnetic resonance Imaging (MRI) for the description of the abnormalities seen in Allergic BronchoPulmonary Aspergillosis (ABPA).

DETAILED DESCRIPTION:
The ABPA is responsible for pulmonary exacerbations in chronic bronchial diseases. The treatment of ABPA consists in systemic corticosteroids and anti fungal therapy, which can have severe side effects. The diagnosis is difficult, based on several but non-specific characteristics. One of the radiologic abnormalities on CTscan could be more specific : high attenuation in impacted mucus, but this sign is found in about 30% of cases. Recent articles and investigators experience seem to demonstrate that MRI could provide an interesting tool for ABPA diagnosis, studying the signal of bronchial impactions. The aim of the study is to describe the MRI characteristics of patients with ABPA and compare the results with those obtained by CTscan, and in order to determine if there is a specific signal of impaction in ABPA.

ELIGIBILITY:
Inclusion Criteria:

* study patients have a diagnosis of ABPA
* control patients have severe asthma
* All the patients are ≥ 18 years old, have social security care, signature of consent form

Exclusion Criteria:

* cystic fibrosis
* other type of aspergilloses
* contraindication for MRI
* woman without effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Concordance between chest CT scan and MRI for bronchial and pulmonary signs of ABPA (bronchiectases, infiltrates, impactions) | Day 0
  Measured by a kappa test

CONTACTS AND LOCATIONS:
Overall Officials: Julie MACEY, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, France